CLINICAL TRIAL: NCT03002181
Title: The Effect of Pain Neurophysiology Education on Sport Therapy Students Knowledge, Attitudes and Clinical Behaviour Towards Athletes With Chronic Pain: a Randomised Control Trial
Brief Title: Pain Neurophysiology Education for Sport Therapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Neil Maguire, Graduate Tutor, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PNE Edu
Record Dates: First submitted 2016-11-18; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Knowledge; Attitude; Behavior
MeSH Terms: conditions — Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PNE group (Experimental): Pain neurophysiology education group.
  Interventions: Other: Education
- Red Flag group (Experimental): Red Flags education group.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — 70 minute education session.

SUMMARY:
The effect of a 70 minute Pain Neurophysiology Education session on Sport Therapy Students Knowledge, Attitudes and Clinical Behaviour Towards Athletes With Chronic Pain

DETAILED DESCRIPTION:
This single-blind, randomised control trial aims to investigate the effect of a brief 70 minute Pain Neurophysiology Education session on sport therapy students knowledge, attitudes and clinical behaviour towards athletes with chronic pain. Participants will be selected from first year undergraduate and postgraduate sport therapy cohorts. Random number generator will assign participants into two subgroups. Group 1 will receive a control education on clinical 'red flags'. Red flags are questions that are routinely asked by therapists in clinical practice to screen for sinister pathology. Group 2 will receive education called 'Pain Neurophysiology Education' (taken from the Explain Pain publication). This mode of education uses the neurophysiology of pain to explain the experience, and has been used as an educational tool for patient, healthcare practitioners and students alike. Data collection (completion of three questionnaires) will take place immediately prior, and immediately after each education session.

The change in these outcomes pre and post intervention will subsequently be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* 1st year undergraduate sport therapy students
* 1st year postgraduate, pre-registration sport therapy students
* Enrolled at Teesside University, UK.

Exclusion Criteria:

* Previous detailed pain education on either PNE or Red Flags.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain Neurophysiology Quiz. (knowledge) | Outcome measure assessed IMMEDIATELY post intervention, on the same day. NO FOLLOW UP.
  A 13 point validated questionnaire assessing participant knowledge of contemporary pain knowledge.
The Health Care Pain Attitudes and Impairment Relationship Scale. (attitudes) | Outcome measure assessed IMMEDIATELY post intervention, on the same day. NO FOLLOW UP.
  A 13 item validated likert-scale questionnaire to measure health care professionals attitudes towards the ability of patients with pain to function despite their pain.
Clinical Vignette. (clinical recommendations) | Outcome measure assessed IMMEDIATELY post intervention, on the same day. NO FOLLOW UP.
  A case vignette is a validated proxy measure of clinical behaviour, and is assessed by multiple choice recommendations following a case scenario. This recommendations are weighted as either 'appropriate' or 'inappropriate' based on current clinical guidelines.

IPD SHARING:
Plan to Share IPD: No
No identifiable data was used in the current study